CLINICAL TRIAL: NCT06593119
Title: Tailoring a Telemedicine Hypertension Management Intervention for Black Patients
Brief Title: Tailoring TM-HTN Intervention for Black Patients
Acronym: TM-HTN
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00116281; 11773 (Other Grant/Funding Number: NHLBI)
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Hypertension
Keywords: Telemedicine; socially disadvantaged; African American or Black patients
MeSH Terms: conditions — Hypertension | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: 60 patients total (30 in the TM-HTN intervention group, 30 in the control group).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telemedicine management of Hypertension intervention group (Experimental): BP monitor and telehealth application Home BP monitoring Pharmacotherapy Telemedicine-based self-management support Additional support in-person training
  Interventions: Behavioral: Telemedicine management of Hypertension
- control group (Placebo Comparator): This includes usual clinic based Hypertension care using routinely available clinic resources (e.g., community health worker, social worker). Clinicians can offer self-management support (e.g., dietician referral) or recommend a home BP monitor. These activities mirror current primary care practice.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Telemedicine management of Hypertension — TM-HTN intervention includes tailored and frequent self-management support, home blood pressure monitoring, pharmacotherapy, and as-needed assistance for health-related social needs provided by pharmacists, nurses, community health workers, and social workers. This will be compared with usual care
  Other Names: TM-HTN
  Arms: Telemedicine management of Hypertension intervention group
Behavioral: Usual Care — This includes usual clinic based HTN care using routinely available clinic resources (e.g., community health worker, social worker). Clinicians can offer self-management support (e.g., dietician referral) or recommend a home BP monitor. These activities mirror current primary care practice.
  Other Names: Control Group
  Arms: control group

SUMMARY:
Current clinic-based hypertension (HTN) management models have several limitations, resulting in episodic care that does not adequately support patients' self-care skills, and fails to achieve blood pressure (BP) control.

DETAILED DESCRIPTION:
Telemedicine management of HTN (TM-HTN) can augment and overcome challenges by allowing more support for patients' HTN self-care skills, providing multiple home Blood Pressure values and overcoming failure to appropriately intensify treatment. TM-HTN consists of 1) home BP monitoring, 2) home BP based pharmacotherapy, and 3) telemedicine-based self-management support.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be African American or Black
* experiencing socially disadvantage
* Patients with systolic Blood Pressure ≥140 mmHg on their last two clinic visits and baseline systolic BP >130 mmHg using the mean of two research BP values measured by trained staff
* Subjects must be on stable Blood Pressure medications for the preceding 6 weeks

Exclusion Criteria:

* Unable to read or speak English
* diminished ability to measure home Blood Pressure
* chronic kidney disease ≥stage 4
* persistent/chronic atrial fibrillation
* severe hypertension >180/110 mmHg
* acute health changes in past 3 months increasing chance of Blood Pressure instability
* terminal illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-08 (Estimated); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who are screened | Month 6
  Proportion of patients who are screened
Proportion of patients who are eligible | Month 6
  Proportion of patients who are eligible
Proportion of patients who agree to participate | Month 6
  Proportion of patients who agree to participate
Proportion of patients who decline | Month 6
  Proportion of patients who decline
Number of staff needed and time spent for intervention | Month 6
  staff training, technical support, troubleshooting
Proportion of completed self-measurement of Blood Pressure at home | Month 6
  Proportion of completed self-measurement of BP at home
Proportion of completed self-management contacts. | Month 6
  Proportion of completed self-management contacts.

SECONDARY OUTCOMES:
Change in Blood Pressure | Month 6
  Effect size for BP change at 6-months (both arms)
Medication adherence | Month 6
  Medication adherence using the Proportion of Days Covered and Domains of Subjective Extent of Nonadherence Measure (both arms)
Feasibility of Intervention Measure [FIM] | Month 6
  measured on a 5-point Likert scale - 'excellent', 'good', 'fair' or 'poor' - higher scores denotes better feasibility
Acceptability of Intervention Measure [AIM] | Month 6
  Items are measured on a 5-point Likert scale (Completely Disagree-Completely Agree)
Intervention Appropriateness Measure [IAM] | Month 6
  The IAM uses a 5-point Likert scale, with scores ranging from "Completely Disagree" to "Completely Agree". The mean of the scores is calculated to determine the overall score.
Patient Assessment of Chronic Illness Care [PACIC] | Month 6
  The Patient Assessment of Chronic Illness Care (PACIC) is scored by averaging the responses to all 20 items on the scale. The score ranges from 1 to 5, with higher scores indicating that patients feel more involved in their care and self-management.
Organizational Readiness for Implementing Change [ORIC] | Month 6
  Organizational Readiness for Implementing Change (ORIC) is a 12-item instrument used to determine how well employees at an organization feel they can implement the change in processes required by a proposed intervention. Each item includes a Likert scale from 1 (Disagree) to 5 (Agree) - The range of each scale is -10 through 0 to +10. A negative scale score reflects an overall disagreement with items measuring the stage of change, whereas a positive score represents overall agreement.

OTHER OUTCOMES:
Number of clinic, urgent care and emergency department visits | Month 6
  Number of clinic, urgent care and emergency department visits from Electronic Medical Records (both arms).
Patient self-reported home BP monitor use | Month 6
  Patient self-reported home BP monitor use and self-management referrals from EMR (usual care group only).
Reasons for patient contact | Month 6
  Reasons for patient contact (scheduled, unscheduled calls [e.g., technical, intervention or safety related]) (TM-HTN arm only)
patients with resistant hypertension | Month 6
  Subgroup analysis in patients with resistant hypertension

CONTACTS AND LOCATIONS:
Overall Officials: Yashashwi Pokharel, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No